CLINICAL TRIAL: NCT01098994
Title: Pilot and Feasibility Study for a Pharmacogenomic Trial in Type 1 Diabetes
Brief Title: Haptoglobin Phenotype, Vitamin E and High-density Lipoprotein (HDL) Function in Type 1 Diabetes
Acronym: HAP-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Tina Costacou, Assistant Professor of Epidemiology, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-10-CT-12; 1-10-CT-12 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2010-02-24; First posted 2010-04-06 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Type 1 Diabetes; Heart Disease
Keywords: Type 1 diabetes; Haptoglobin genotype; HDL function; Heart disease; Feasibility of clinical trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Heart Diseases | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Haptoglobin 1/1 (Other): Individuals with type 1 diabetes and the Haptoglobin 1/1 phenotype
  Interventions: Dietary Supplement: Vitamin E; Other: Dummy pills
- Haptoglobin 2/1 (Other): Individuals with type 1 diabetes and the Haptoglobin 2/1 phenotype
  Interventions: Dietary Supplement: Vitamin E; Other: Dummy pills
- Haptoglobin 2/2 (Other): Individuals with type 1 diabetes and the Haptoglobin 2/2 phenotype
  Interventions: Dietary Supplement: Vitamin E; Other: Dummy pills

INTERVENTIONS:
Dietary Supplement: Vitamin E — Daily administration of 400 IU natural d-alpha tocopherol acetate for 8 weeks
  Other Names: Natural d-alpha tocopherol acetate
Other: Dummy pills — Daily placebo administration for 8 weeks
  Other Names: Placebo, inactive pills

SUMMARY:
The purpose of the study is to determine whether the function of the good cholesterol (HDL cholesterol) as well as its subfractions (via NMR spectroscopy) is altered among people with type 1 diabetes and a variation in the Haptoglobin gene and to evaluate whether vitamin E supplements may improve this function.

DETAILED DESCRIPTION:
Persons with type 1 diabetes are at a much greater risk for heart disease compared to the general population. Among individuals with diabetes, those with a specific variation in a genetic marker called Haptoglobin (approximately 43% of persons with type 1 diabetes) are at even greater risk compared to those not carrying this genetic variation. A genetic marker or a "gene" is information inherited from parents (a blueprint) about the structure and functions of cells in the body that make up the color of our hair and eyes and may influence the way our bodies respond to certain stimuli such as an illness, or infection.

In this project we are seeking to understand what some of the mechanisms may be that put persons with type 1 diabetes and this variation in the Haptoglobin gene at greater risk for heart disease. Specifically, we will assess whether this gene variant affects the function of the good cholesterol (HDL cholesterol) and its subfractions (via NMR spectroscopy), which is thought to help against heart disease development. We also seek to evaluate whether vitamin E supplements may improve this function. If results indicate that vitamin E is beneficial and improves the function of HDL cholesterol, the next question to be answered would be whether vitamin E would also help reduce the risk of heart disease itself in these persons. To answer the latter, a large clinical trial would have to take place. In this research project we will therefore also evaluate whether such a trial would be feasible and whether individuals with type 1 diabetes would be interested in participating in a long, 4-5 year, clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 1 diabetes residing in the Pittsburgh, PA area (members of the Allegheny Count or Children's Hospital of Pittsburgh/Epidemiology of Diabetes Complications Registries)
* 30 years old or older
* with diabetes duration greater than 10 years or less than 10 years but with a history of heart disease

Exclusion Criteria:

* Allergy to vitamin E
* Stroke, MI within the past 6 months
* Unwillingness/inability to limit antioxidant supplement use to study-provided supplements

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Demonstrate the presence of HDL dysfunction among individuals with the Haptoglobin 2/1 and 2/2 compared to those with the Hp 1/1 phenotype and improvement in HDL dysfunction with natural d-α-tocopherol supplementation | 6 months
  HDL-associated lipid peroxides, HDL function (based on its ability to promote cholesterol efflux from macrophages), HDL antioxidant and anti-inflammatory activities; NMR lipoprotein subfractions will be assessed

SECONDARY OUTCOMES:
Feasibility of recruitment of individuals with type 1 diabetes for a randomized clinical trial | 1 year
  Members of two registries (ACR and CHP/EDC) residing within 100 miles or 2.5 hours driving distance from Pittsburgh, Pennsylvania will be contacted and interest for participation in a trial will be assessed as part of the original registry's follow-up. Investigators will contact those interested, explain the study aims and scope, and further assess willingness and eligibility for participation in a clinical trial.
Assessment of adherence to the clinical trial study protocol in a random sample of individuals with type 1 diabetes recruited from the ACR and CHP/EDC Diabetes Registries | 6 months
  Protocol adherence will be evaluated by clinic attendance, pill count and by comparison of plasma α-tocopherol concentrations at baseline with plasma levels after vitamin E supplementation or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Costacou, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Diabetes and Lipid Research Clinic, Pittsburgh, Pennsylvania, United States